CLINICAL TRIAL: NCT00036452
Title: A Randomized, Phase II, Open Label Study to Compare Twice Daily and Once Daily Potent Antiretroviral Therapy and to Compare Self-Administered Therapy and Therapy Administered Under Direct Observation
Brief Title: A Study to Compare Anti-HIV Drugs Given Twice a Day or Once a Day, With or Without Direct Observation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A5073; 10073 (Registry Identifier: DAIDS ES); ACTG A5073; AACTG A5073
Record Dates: First submitted 2002-05-10; First posted 2002-05-13 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Lopinavir; HIV-1; Drug Administration Schedule; Stavudine; HIV Protease Inhibitors; Ritonavir; Reverse Transcriptase Inhibitors; Self Care; Viral Load; Emtricitabine; Directly Observed Therapy; Tenofovir Disoproxil Fumarate; Treatment Naive
MeSH Terms: conditions — HIV Infections; Directly Observed Therapy | interventions — Lopinavir; Emtricitabine; Stavudine; Tenofovir

INTERVENTIONS:
Drug: lopinavir/ritonavir
Drug: emtricitabine
Drug: stavudine
Drug: tenofovir DF

SUMMARY:
Anti-HIV drug therapy works best when the drugs are taken exactly as prescribed by a doctor. Because anti-HIV therapy often involves multiple drugs, some people have difficulty taking them all correctly. The easier it is to take anti-HIV drugs, the more likely people will take them as prescribed and get the best results. This study will see if people are more successful in taking anti-HIV drugs once a day or twice a day. It also will determine if having a health care professional oversee each weekday dose helps people control their HIV infection. The study will compare taking a three-drug combination twice a day versus taking a three-drug combination just once a day. The study will also compare patients taking the drugs on their own to patients taking the drugs in the presence of a clinical worker. Viral load (amount of HIV in the blood) and drug side effects will be measured.

DETAILED DESCRIPTION:
While many factors contribute to the success or failure of antiretroviral therapy for HIV, among the most important are factors that influence adherence to a treatment regimen, such as duration of therapy, dosing frequency, pill burden, side effects, and patient behaviors. Inconsistent adherence or nonadherence to antiretroviral therapy can result in suboptimal drug exposure. Suboptimal drug exposure can, in turn, impact short- and long-term patient outcomes by increasing the likelihood of drug resistant HIV mutants and subsequent virologic and clinical failure. It is therefore essential to design treatment regimens that promote long-term adherence to potent antiretroviral therapy. This study will evaluate the relative contribution of reduced-frequency dosing and directly observed therapy on the magnitude and durability of virologic suppression in patients treated with potent antiretroviral therapy.

Patients will be randomly assigned to one of three study arms. Arms A, B, and C receive the same daily dosage of lopinavir/ritonavir (LPV/r), emtricitabine (FTC), and stavudine extended release (d4T XR) or tenofovir DF (TDF). In Arm A, drugs are self-administered for 48 weeks; LPV/r is taken twice daily and FTC and d4T XR or TDF once daily. In Arm B, all drugs are self-administered once daily for 48 weeks. In Arm C, drugs are taken once a day under directly observed therapy during Weeks 0-24, and then by self-administration during Weeks 25-48. Adherence to the regimen is measured using an electronic drug monitoring system. Viral load, CD4 and CD8 T cell responses, population pharmacokinetics, and quality of life indicators are measured throughout the study. The tolerability and safety of the treatment regimens are also monitored.

ELIGIBILITY:
Inclusion Criteria

* HIV infection
* Age 13 years or older and have written consent of guardian if under 18
* Weigh at least 88 pounds
* Viral load of 2000 copies/ml or more within 90 days before study entry
* Have not taken anti-HIV drugs for more than 7 days
* Agree to use acceptable methods of contraception during the study and for 1 month after stopping the study drugs

Exclusion Criteria

* Pregnant or breastfeeding
* In jail
* Sensitive or allergic to any part of the study drugs
* Treated with acute systemic therapy for a serious infection or other serious medical illness within 7 days prior to study entry, unless the participant has completed 7 days of therapy and is clinically stable
* Recent serious illness, including pancreatitis or peripheral neuropathy
* Alcohol or illicit drug abuse
* Taken any of the following within 14 days before study entry: investigational drugs, anti-HIV vaccines, drugs that may cause pancreatitis or peripheral neuropathy, or drugs that are associated with CYP3A
* Treated for cancer (not including minimal Kaposi's sarcoma) within 30 days before study entry
* History of mental illness that might interfere with the study

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 402 (Actual)
Dates: Study Completion 2006-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donna Mildvan, MD, Study Chair — Beth Israel Medical Center; Charles Flexner, MD, Study Chair — Johns Hopkins University Hospital
Locations (29):
- United States (27):
  - USC CRS, Los Angeles, California
  - Univ. of California Davis Med. Ctr., ACTU, Sacramento, California
  - Ucsd, Avrc Crs, San Diego, California
  - University of Colorado Hospital CRS, Aurora, Colorado
  - Univ. of Miami AIDS CRS, Miami, Florida
  - Univ. of Hawaii at Manoa, Leahi Hosp., Honolulu, Hawaii
  - Indiana Univ. School of Medicine, Infectious Disease Research Clinic, Indianapolis, Indiana
  - IHV Baltimore Treatment CRS, Baltimore, Maryland
  - Johns Hopkins Adult AIDS CRS, Baltimore, Maryland
  - SSTAR, Family Healthcare Ctr., Fall River, Massachusetts
  - University of Minnesota, ACTU, Minneapolis, Minnesota
  - Beth Israel Med. Ctr., ACTU, New York, New York
  - NY Univ. HIV/AIDS CRS, New York, New York
  - Univ. of Rochester ACTG CRS, Rochester, New York
  - AIDS Care CRS, Rochester, New York
  - McCree McCuller Wellness Ctr. at the Connection, Infectious Disease Unit, Rochester, New York
  - Unc Aids Crs, Chapel Hill, North Carolina
  - Regional Center for Infectious Disease, Wendover Medical Center CRS, Greensboro, North Carolina
  - Wake County Health and Human Services CRS, Raleigh, North Carolina
  - Univ. of Cincinnati CRS, Cincinnati, Ohio
  - MetroHealth CRS, Cleveland, Ohio
  - The Ohio State Univ. AIDS CRS, Columbus, Ohio
  - Hosp. of the Univ. of Pennsylvania CRS, Philadelphia, Pennsylvania
  - Pitt CRS, Pittsburgh, Pennsylvania
  - The Miriam Hosp. ACTG CRS, Providence, Rhode Island
  - Vanderbilt Therapeutics CRS, Nashville, Tennessee
  - University of Washington AIDS CRS, Seattle, Washington
- Puerto Rico-AIDS CRS, San Juan, Puerto Rico
- Wits HIV CRS, Johannesburg, Gauteng, South Africa

REFERENCES:
- [Background] Liu H, Golin CE, Miller LG, Hays RD, Beck CK, Sanandaji S, Christian J, Maldonado T, Duran D, Kaplan AH, Wenger NS. A comparison study of multiple measures of adherence to HIV protease inhibitors. Ann Intern Med. 2001 May 15;134(10):968-77. doi: 10.7326/0003-4819-134-10-200105150-00011. PMID 11352698
- [Background] Paterson DL, Swindells S, Mohr J, Brester M, Vergis EN, Squier C, Wagener MM, Singh N. Adherence to protease inhibitor therapy and outcomes in patients with HIV infection. Ann Intern Med. 2000 Jul 4;133(1):21-30. doi: 10.7326/0003-4819-133-1-200007040-00004. PMID 10877736
- [Background] Volmink J, Matchaba P, Garner P. Directly observed therapy and treatment adherence. Lancet. 2000 Apr 15;355(9212):1345-50. doi: 10.1016/S0140-6736(00)02124-3. PMID 10776760
- [Background] Bangsberg DR, Mundy LM, Tulsky JP. Expanding directly observed therapy: tuberculosis to human immunodeficiency virus. Am J Med. 2001 Jun 1;110(8):664-6. doi: 10.1016/s0002-9343(01)00729-x. No abstract available. PMID 11382379
- [Background] Kirkland LR, Fischl MA, Tashima KT, Paar D, Gensler T, Graham NM, Gao H, Rosenzweig JR, McClernon DR, Pittman G, Hessenthaler SM, Hernandez JE; NZTA4007 Study Team. Response to lamivudine-zidovudine plus abacavir twice daily in antiretroviral-naive, incarcerated patients with HIV infection taking directly observed treatment. Clin Infect Dis. 2002 Feb 15;34(4):511-8. doi: 10.1086/338400. Epub 2002 Jan 4. PMID 11797179
- [Result] Gross R, Tierney C, Andrade A, Lalama C, Rosenkranz S, Eshleman SH, Flanigan T, Santana J, Salomon N, Reisler R, Wiggins I, Hogg E, Flexner C, Mildvan D; AIDS Clinical Trials Group A5073 Study Team. Modified directly observed antiretroviral therapy compared with self-administered therapy in treatment-naive HIV-1-infected patients: a randomized trial. Arch Intern Med. 2009 Jul 13;169(13):1224-32. doi: 10.1001/archinternmed.2009.172. PMID 19597072
- [Result] Flexner C, Tierney C, Gross R, Andrade A, Lalama C, Eshleman SH, Aberg J, Sanne I, Parsons T, Kashuba A, Rosenkranz SL, Kmack A, Ferguson E, Dehlinger M, Mildvan D; ACTG A5073 Study Team. Comparison of once-daily versus twice-daily combination antiretroviral therapy in treatment-naive patients: results of AIDS clinical trials group (ACTG) A5073, a 48-week randomized controlled trial. Clin Infect Dis. 2010 Apr 1;50(7):1041-52. doi: 10.1086/651118. PMID 20192725